CLINICAL TRIAL: NCT00288353
Title: Estimating and Reducing the Cardiovascular Risk of Patients With Schizophrenia Drugs From Lipid Measures and Ischemic Electrocardiographic Changes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: unable to secure additional funding
Sponsor: Northwestern University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 050943; NARSAD
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: schizophrenia; schizoaffective disorder; bipolar disorder; metabolic syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Metabolic Syndrome | interventions — Aripiprazole; ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): aripiprazole (Abilify)
  Interventions: Drug: aripiprazole (Abilify)
- 2 (Active Comparator): ziprasidone (Geodon)
  Interventions: Drug: ziprasidone (Geodon)

INTERVENTIONS:
Drug: aripiprazole (Abilify) — active drug given daily as per package insert according to standard clinical care for twelve month duration of study. Subject will be switched from current antipsychotic to this drug or other randomized study medication.
  Arms: 1
Drug: ziprasidone (Geodon) — active medication will be given daily as per package insert according to standard clinical care for the twelve month duration of the study. Subject will be switched from current antipsychotic medication to this medication or the other randomized medication.
  Arms: 2

SUMMARY:
The primary goal of this study is to examine the triglyceride/high-density lipoprotein (TG/HDL) ratio and the ischemic EKG changes in patients with schizophrenia, schizoaffective disorder or bipolar disorder.

DETAILED DESCRIPTION:
The primary goal of this study is to examine the triglyceride/high-density lipoprotein (TG/HDL) ratio and the ischemic EKG changes in patients with schizophrenia, schizoaffective disorder or bipolar disorder. The secondary goal is to identify those subjects in the top tertile for the highest risk of ischemic heart disease (IHD) as defined by TG/HDL ratios (>>3.5) and ischemic EKG changes with and without clinical ischemia, e.g. angina and to see if these risk factors can be reduced or reversed by a change of antipsychotic medication, dietary counseling, enrollment into available exercise groups, etc.

ELIGIBILITY:
Inclusion criteria

To be eligible, a patient must :

* Be male or female, between 18-65.
* Have a diagnosis of schizophrenia, schizoaffective disorder or bipolar disorder according to Diagnostic and Statistical Manual (DSM-IV) criteria
* Have TG/HDL ratios (>>3.5) and ischemic EKG changes with and without clinical ischemia, e.g. angina
* Be treated for a minimum of six months with one of six oral antipsychotic medications: clozapine, haloperidol, olanzapine, quetiapine, risperidone and ziprasidone
* Be willing to change current antipsychotic medication to that chosen by the principal investigator
* Have a history of compliance with the above medication
* Be Medicaid eligible or maintain insurance covering requested lab procedures
* Be able to provide written informed consent.

Exclusion criteria

A patient will be considered ineligible if he/she:

* Has a diagnosis other than schizophrenia, schizoaffective disorder or bipolar disorder with psychotic features according to DSM-IV criteria.
* Has a history of noncompliance with prescribed psychiatric medications
* Has a TG/HDL ratio < 3.5 on current medication
* Is uninsured or is unable to self-pay potential costs of required lab procedures not covered by insurance.
* Is unable to provide written informed consent.
* (Females only) Is pregnant, lactating or plans to become pregnant during study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tianlai Tang, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole (Abilify): aripiprazole (Abilify): active drug given daily as per package insert according to standard clinical care for the twelve-month duration of study. Subject will be switched from current antipsychotic to this drug or other randomized study medication.
- Ziprasidone (Geodon): ziprasidone (Geodon): active medication will be given daily as per package insert according to standard clinical care for the twelve-month duration of the study. Subject will be switched from current antipsychotic medication to this medication or the other randomized medication.
Period: Overall Study
Arm/Group | Aripiprazole (Abilify) | Ziprasidone (Geodon)
Started | 25 | 23
Completed | 18 | 16
Not Completed | 7 | 7
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole (Abilify) | Ziprasidone (Geodon) | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (8.5) | 45.5 (9.4) | 44.9 (8.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Self-Reported Gender: Male | 9 | 10 | 19
  Self-Reported Gender: Female | 16 | 13 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hypertension, number [Count of Participants; unit: Participants]
  Participants with hypertension | 13 | 3 | 16
  Participants without hypertension | 12 | 20 | 32
Type 2 Diabetes, number [Count of Participants; unit: Participants]
  Participants with Type 2 Diabetes | 4 | 5 | 9
  Participants without Type 2 Diabetes | 21 | 18 | 39
Diagnosis of schizophrenia (SCH) and schizoaffective disorder (SCHAF) or bipolar disorder number [Count of Participants; unit: Participants]
  schizophrenia (SCH) or schizoaffective disorder (SCHAF) | 14 | 9 | 23
  bipolar disorder | 11 | 14 | 25
Positive and Negative Syndrome Scale (PANSS) Total Score [Least Squares Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale (PANSS) is a 30-item questionnaire for assessing severity of schizophrenia symptoms. The PANSS is divided into three subscales: positive symptoms, negative symptoms, and cognitive. Each item is rated on a 7-point scale, ranging from absent to extreme. Therefore, the minimum possible score of 0 and maximum possible score is 210, but those scores may never be seen in a practical setting. If the score reduces over time that indicates improvement of the symptoms.
  units on a scale | 61.3 (2.2) | 61.0 (2.2) | 61.15 (2.2)
Positive and Negative Syndrome Scale (PANSS) Positive Score [Least Squares Mean (Standard Deviation); unit: units on a scale] — Positive and Negative Syndrome Scale (PANSS) Positive scale; the scale consists of a sum of 7 items, so the score can range from 0 - 49. Improvement means lower scores over time
  units on a scale | 14.2 (0.7) | 14.2 (0.7) | 14.2 (0.7)
Positive and Negative Syndrome Scale (PANSS) Negative Score [Least Squares Mean (Standard Deviation); unit: units on a scale] — Positive and Negative Syndrome Scale (PANSS) Negative scale; the scale consists of a sum of 7 items, so the score can range from 0 - 49. Improvement means lower scores over time
  units on a scale | 15.3 (0.7) | 15.2 (0.6) | 15.25 (0.65)
Positive and Negative Syndrome Scale (PANSS) Cognitive Score [Least Squares Mean (Standard Deviation); unit: units on a scale] — Positive and Negative Syndrome Scale (PANSS) Positive scale; the scale consists of a sum of 16 items, so the score can range from 0 - 112. Improvement means lower scores over time
  units on a scale | 6.7 (0.4) | 6.6 (0.4) | 6.65 (0.4)
Drug taken prior to enrollment [Count of Participants; unit: Participants]
  Olazapine | 4 | 4 | 8
  Quetiapine | 10 | 9 | 19
  Risperidone | 8 | 7 | 15
  Typical neuroleptics | 2 | 1 | 3
  Mood stabilizer only | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Triglyceride/High-density Lipoprotein (TG/HDL) Ratio
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: (mg/dL)/(mg/dL)
Arm/Group | Aripiprazole (Abilify) | Ziprasidone (Geodon)
Number analyzed (Participants) | 25 | 23
(mg/dL)/(mg/dL)
  Baseline | 8.1 (0.7) | 8.2 (0.6)
  6 weeks | 4.9 (0.7) | 4.7 (0.7)
  12 weeks | 4.8 (0.7) | 5.6 (0.7)
  24 weeks | 5.7 (0.9) | 5.2 (0.7)

2. Secondary Outcome: Weight
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: lbs
Arm/Group | Aripiprazole (Abilify) | Ziprasidone (Geodon)
Number analyzed (Participants) | 25 | 23
lbs
  Baseline | 216.8 (2.4) | 216.7 (2.2)
  6 weeks | 211.8 (2.5) | 208.8 (2.3)
  12 weeks | 211.2 (2.6) | 209.4 (2.5)
  24 weeks | 210.9 (3.0) | 207.1 (2.5)

3. Secondary Outcome: Body Mass Index (BMI)
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Aripiprazole (Abilify) | Ziprasidone (Geodon)
Number analyzed (Participants) | 25 | 23
kg/m^2
  Baseline | 35.5 (0.4) | 35.5 (0.4)
  6 weeks | 34.7 (0.4) | 34.1 (0.4)
  12 weeks | 34.6 (0.4) | 34.3 (0.5)
  24 weeks | 34.4 (0.5) | 33.9 (0.4)

4. Secondary Outcome: Cholesterol
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/DL
Arm/Group | Aripiprazole (Abilify) | Ziprasidone (Geodon)
Number analyzed (Participants) | 25 | 23
mg/DL
  Baseline | 210.4 (8.8) | 211.7 (7.9)
  6 Weeks | 193.0 (9.1) | 203.7 (8.4)
  12 Weeks | 209.2 (9.4) | 193.2 (9.0)
  24 Weeks | 197.7 (10.3) | 85.9 (9.3)

5. Secondary Outcome: High-Density Lipoprotein (HDL)
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Aripiprazole (Abilify) | Ziprasidone (Geodon)
Number analyzed (Participants) | 25 | 23
mg/dL
  Baseline | 39.7 (1.6) | 38.4 (1.5)
  6 Weeks | 42.0 (1.7) | 45.0 (1.6)
  12 Weeks | 43.5 (1.8) | 45.0 (1.7)
  24 Weeks | 43.5 (2.1) | 42.3 (1.8)

6. Secondary Outcome: Triglyceride (TG)
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Aripiprazole (Abilify) | Ziprasidone (Geodon)
Number analyzed (Participants) | 25 | 23
mg/dL
  Baseline | 306.1 (27.1) | 303.5 (25.1)
  6 Weeks | 204.3 (29.7) | 202.5 (27.1)
  12 Weeks | 198.8 (29.7) | 228.5 (28.8)
  24 Weeks | 238.7 (36.3) | 208.1 (30.8)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Arm/Group | Aripiprazole (Abilify) | Ziprasidone (Geodon)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No